CLINICAL TRIAL: NCT00748709
Title: An Open Label Phase II Trial of BIBW 2992 (Afatinib) in Genetically Pre-screened Cancers With EGFR and/or HER2 Gene Amplification or EFGR Activating Mutations.
Brief Title: Phase II Trial of BIBW 2992 (Afatinib) in Genetically Pre-screened Cancers With EGFR and/or HER2 Gene Amplification.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1200.26
Record Dates: First submitted 2008-09-08; First posted 2008-09-09 (Estimated); Results first posted 2013-10-14 (Estimated); Last update posted 2025-02-11 (Actual); Status verified 2025-01

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — Afatinib

ARMS (1):
- BIBW 2992 (Afatinib) (Experimental): BIBW 2992 (Afatinib) for patients FISH positive for/or harboring EGFR or HER2 Mutation
  Interventions: Drug: BIBW 2992 (Afatinib)

INTERVENTIONS:
Drug: BIBW 2992 (Afatinib) — BIBW 2992 (Afatininb) for patients FISH positive for/or harboring EGFR or HER2 Mutation

SUMMARY:
This is a Phase II open-label exploratory trial of BIBW 2992 administered to patients with tumors of various histologies found to possess EGFR and/or HER2 gene amplification, or EGFR activating mutations.

ELIGIBILITY:
Inclusion criteria:

There are 2 Steps in the screening process:

Step 1 Inclusion criteria for pre-screening:

1. Histologically confirmed diagnosis of advanced cancer of one of the following four tumor type categories:

   Category 1, Gastric, GE junction, or Esophageal cancer Category 2, Biliary or gallbladder cancer Category 3, TCC urothelial tract, and Category 4, Gynecological cancers
2. Measurable disease by RECIST criteria.
3. Willingness and ability to give written informed consents consistent with ICHGCP guidelines.
4. Life expectancy of at least three (3) months.
5. Eastern Cooperative Oncology Group performance score 0, 1 or 2.
6. Age >18 years.

Step 2 Inclusion criteria for enrollment:

Patients who have tested positive for FISH and are considered candidate for this trial must meet all of the following inclusion criteria:

1. Histologically confirmed diagnosis of advanced cancer of one of the following four tumor type categories:

   Category 1, Gastric, GE junction, or Esophageal cancer Category 2, Biliary or gallbladder cancer Category 3, TCC urothelial tract, and Category 4, Gynecological cancers
2. Documented failure to respond or progression of underlying cancer after at least one line of prior chemotherapy.
3. EGFR and/or HER2 gene amplification by FISH testing or patients with tumors that harbor known activating EGFR mutations.
4. Measurable disease by RECIST criteria.
5. Willingness and ability to give written informed consents consistent with ICH-GCP guidelines.
6. Life expectancy of at least three (3) months.
7. Eastern Cooperative Oncology Group performance score 0, 1 or 2.
8. Age >18 years.

Exclusion criteria:

1. Prior treatment with gefitinib, erlotinib, lapatinib and/or other EGFR TKIs.
2. Treatment with cytotoxic anti-cancer-therapies or investigational drugs during the last four weeks prior to the first treatment with the trial drug. (a shorter duration may be considered for patients treated with oral, non cytotoxic drugs on an individual basis and upon discussion between the principal investigator and sponsor)
3. Inability to take BIBW 2992 by mouth (BIBW 2992 may not be crushed or administered via Gastrostomy-tube)
4. Chronic diarrhea or other gastrointestinal disorders that may interfere with the absorption of the trial drug.
5. History of other malignancies unless free of disease for at least 3 years (except for appropriately treated superficial non-melanoma skin cancer and surgically cured cervical cancer in situ).
6. History or presence of clinically relevant cardiovascular abnormalities such as uncontrolled hypertension, congestive heart failure NYHA classification of 3, unstable angina or poorly controlled arrhythmia. Myocardial infarction within 6 months prior to randomization.
7. Resting left ventricular ejection fraction <50% OR below the institution's lower limit of normal (if the institutions lower limit is above 50%), measured by MUGA scan or echocardiogram.
8. Active infectious disease
9. Serious illness, concomitant non-oncological disease or mental problems considered by the investigator to be incompatible with participation in this trial.
10. Active/symptomatic brain metastases. Patients with a history of treated brain metastases must have stable or normal brain MRI scan at screening and be at least three months post-radiation or surgery for brain metastasis.
11. Absolute Neutrophil Count (ANC) less than 1,000/mm3.
12. Platelet count less than 100,000/mm3.
13. Hemoglobin Level less than 9.0 grams/dl.
14. Total Bilirubin greater than 1.5 mg/dl; higher Total Bilirubin values may be acceptable for patients with known Gilbert¿s disease, approval by the PI and sponsor will be necessary.
15. Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) greater than 3 times the upper limit of normal; or 5 times the upper limit of normal in patients with neoplastic liver involvement.
16. Serum creatinine greater than 1.5 x upper limit of normal for the institution.
17. Patients who are sexually active and unwilling to use simultaneously two medically acceptable method of contraception, one of which being a barrier type method such as condom.
18. Pregnancy or breast-feeding.
19. Patients unable to comply with the protocol
20. Active alcohol and/or substance abuse.
21. Continuation of therapy-related toxicities from prior anti cancer therapies, prior surgery, of CTCAE Grade >=2 at the time of the first administration of the trial drug.
22. Patients with known pre-existing interstitial lung disease.
23. Requirement for treatment with any of the prohibited concomitant medications: additional experimental anti-cancer treatment and/or standard chemotherapy, immunotherapy, hormone treatment or radiotherapy; P-gp inhibitors

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-10-01 (Actual); Primary Completion 2010-11-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (15):
- United States (12):
  - 1200.26.3 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1200.26.11 Boehringer Ingelheim Investigational Site, Denver, Colorado
  - 1200.26.9 Boehringer Ingelheim Investigational Site, Indianapolis, Indiana
  - 1200.26.1 Boehringer Ingelheim Investigational Site, Boston, Massachusetts
  - 1200.26.13 Boehringer Ingelheim Investigational Site, Las Vegas, Nevada
  - 1200.26.4 Boehringer Ingelheim Investigational Site, Albany, New York
  - 1200.26.2 Boehringer Ingelheim Investigational Site, New York, New York
  - 1200.26.7 Boehringer Ingelheim Investigational Site, Kettering, Ohio
  - 1200.26.12 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1200.26.8 Boehringer Ingelheim Investigational Site, Tyler, Texas
  - 1200.26.6 Boehringer Ingelheim Investigational Site, Norfolk, Virginia
  - 1200.26.10 Boehringer Ingelheim Investigational Site, Vancouver, Washington
- Taiwan (3):
  - 1200.26.88603 Boehringer Ingelheim Investigational Site, Tainan
  - 1200.26.88601 Boehringer Ingelheim Investigational Site, Taipei
  - 1200.26.88602 Boehringer Ingelheim Investigational Site, Taoyuan District

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

RESULTS

PARTICIPANT FLOW:
Recruitment Details: "The trial was terminated earlier than planned because of a high screen-failure rate and recruitment challenges that prevented full accrual; no safety or efficacy findings influenced this decision. "
Groups:
- Afatinib 50mg: Patients with genetically pre-screened cancers with EGFR and/or HER2 gene amplification or EGFR activating mutations treated with afatinib 50mg once daily.
Period: Overall Study
Arm/Group | Afatinib 50mg
Started | 20 (Treated)
Completed | 0
Not Completed | 20
Not completed — Progressive disease | 15
Not completed — Drug reducing Toxity | 2
Not completed — Other Adverse Event | 1
Not completed — Withdrawal by Subject | 1
Not completed — Other Reasons | 1

BASELINE CHARACTERISTICS:
Arm/Group | Afatinib 50mg
Number analyzed (Participants) | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 14

OUTCOME MEASURES:

1. Secondary Outcome: Percentage of Participants With Clinical Benefit (CB)
Description: CB was defined as CR, PR or stable disease (SD) and was assessed according to RECIST 1.0 criteria.
Time Frame: Tumour assessments were performed at screening, week 6, week 12, and every 8 weeks till database lock
Population: TS.
Measure: Number; unit: percentage of patients
Arm/Group | Afatinib 50mg
Number analyzed (Participants) | 20
percentage of patients
  With CB | 45.0
  Without CB | 55.0

2. Secondary Outcome: Time to Objective Response (OR)
Description: The time to OR was the duration from the first treatment to the time when the measurement criteria for CR and/or PR were met according to RECIST 1.0 criteria.
Time Frame: Tumour assessments were performed at screening, week 6, week 12, and every 8 weeks till database lock
Population: Trial terminated early, therefore no data summaries produced for time to OR.
Arm/Group | Afatinib 50mg
Number analyzed (Participants) | 0

3. Secondary Outcome: Duration of OR
Description: Duration of OR was measured from the time the criteria for CR or PR (whichever was documented first) were first met until the first date that progressive disease or death was objectively documented.
Time Frame: Tumour assessments were performed at screening, week 6, week 12, and every 8 weeks till database lock.
Population: Trial terminated early, therefore no data summaries produced for duration of OR.
Arm/Group | Afatinib 50mg
Number analyzed (Participants) | 0

4. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the time from the start of treatment to the occurrence of disease progression or death, whichever came first. Disease progression was assessed according to RECIST 1.0 criteria as well as by the investigators assessment, progression date recorded from post trial follow up or start of new anticancer treatment.
Time Frame: Tumour assessments were performed at screening, week 6, week 12, and every 8 weeks till database lock.
Population: Trial terminated early, therefore no data summaries produced for PFS.
Arm/Group | Afatinib 50mg
Number analyzed (Participants) | 0

5. Secondary Outcome: Patients With AEs Resulting in Dose Reduction or Treatment Discontinuation
Description: Patients with adverse events (AEs) resulting in dose reduction or treatment discontinuation
Time Frame: First administration of trial medication until 28 days after last administration of trial medication
Population: TS
Measure: Number; unit: Participants
Arm/Group | Afatinib 50mg
Number analyzed (Participants) | 20
Participants
  With AE leading to drug discontinuation | 5
  With AE leading to dose reduction | 1
  With Treatment held or paused due to AE | 8

6. Secondary Outcome: Maximum CTCAE Grade
Description: Patients with AEs by maximum Common Terminology Criteria for Adverse Events (CTCAE) grade
Time Frame: First administration of trial medication until 28 days after last administration of trial medication
Population: TS
Measure: Number; unit: Participants
Arm/Group | Afatinib 50mg
Number analyzed (Participants) | 20
Participants
  Grade 1 | 2
  Grade 2 | 5
  Grade 3 | 10
  Grade 4 | 0
  Grade 5 | 3

7. Primary Outcome: Percentage of Participants With Objective Response (OR)
Description: OR is defined as the percentage of patients with complete response (CR) or partial response (PR) and was assessed according to the Response Evaluation Criteria in Solid Tumours version 1.0 (RECIST 1.0).
Time Frame: Tumour assessments were performed at screening, week 6, week 12, and every 8 weeks thereafter
Population: Treated Set (TS). TS consisted of all patients who received at least one dose of trial medication.
Measure: Number; unit: percentage of patients
Arm/Group | Afatinib 50mg
Number analyzed (Participants) | 20
percentage of patients | 5.0

8. Secondary Outcome: Pre-dose Concentration of Afatinib in Plasma at Steady State on Day 15 (Cpre,ss,15) for Patients on 50mg on Day 15
Description: Cpre,ss,15 represents the pre-dose concentration of afatinib in plasma at steady state on day 15 for patients on 50mg on day 15.
Time Frame: Day 15
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Afatinib 50mg
Number analyzed (Participants) | 12
ng/mL | 33.2 (80.0)

9. Secondary Outcome: Number of Patients With Diarrhea or Rash
Description: Number of Patients with Diarrhea or Rash
Time Frame: First administration of trial medication until 28 days after last administration of trial medication
Population: TS
Measure: Number; unit: Participants
Arm/Group | Afatinib 50mg
Number analyzed (Participants) | 20
Participants
  AE : Diarrhea | 18
  AE : Rash | 12

ADVERSE EVENTS:
Time Frame: First administration of trial medication until 28 days after last administration of trial medication
Arm/Group | Afatinib 50mg
Serious Adverse Events (participants affected / at risk) | 6/20
Other Adverse Events (participants affected / at risk) | 20/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib 50mg (N=20)
Diarrhoea (Gastrointestinal disorders) | 1
Escherichia bacteraemia (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Female genital tract fistula (Reproductive system and breast disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Afatinib 50mg (N=20)
Anaemia (Blood and lymphatic system disorders) | 4
Constipation (Gastrointestinal disorders) | 3
Diarrhoea (Gastrointestinal disorders) | 17
Dyspepsia (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 7
Stomatitis (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 7
Chest pain (General disorders) | 2
Fatigue (General disorders) | 9
Oedema peripheral (General disorders) | 2
Paronychia (Infections and infestations) | 6
Urinary tract infection (Infections and infestations) | 4
Blood creatinine increased (Investigations) | 2
Weight decreased (Investigations) | 4
Decreased appetite (Metabolism and nutrition disorders) | 11
Dehydration (Metabolism and nutrition disorders) | 4
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 2
Dysgeusia (Nervous system disorders) | 3
Insomnia (Psychiatric disorders) | 4
Haematuria (Renal and urinary disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2
Alopecia (Skin and subcutaneous tissue disorders) | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 6
Dry skin (Skin and subcutaneous tissue disorders) | 4
Pruritus (Skin and subcutaneous tissue disorders) | 4
Rash (Skin and subcutaneous tissue disorders) | 12
Hypotension (Vascular disorders) | 2

LIMITATIONS AND CAVEATS:
Due to early study termination, only data on the primary efficacy endpoint were summarized, no CIs were produced and efficacy and safety results were presented for the overall population rather than by tumor category.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication